CLINICAL TRIAL: NCT01639599
Title: Phase 4 Study of Optimal Dose of Haloperidol
Brief Title: Optimal Haloperidol Dose for Postoperative Nausea and Vomiting Prevention in High-risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, clinical associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: haloperidol
Record Dates: First submitted 2012-07-04; First posted 2012-07-12 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Gynecological Disease
Keywords: non-smoker; female; IV PCA; patient-controlled analgesia
MeSH Terms: conditions — Genital Diseases, Female | interventions — Dexamethasone; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dexamethasone (Placebo Comparator): dexamethasone 5mg iv during anesthesia induction
  Interventions: Drug: Dexamethasone iv injection
- dexamethasone, haloperiol 1mg (Active Comparator): dexamethasone 5mg iv during anesthesia induction & haloperidol 1mg iv 30 min before end of anesthesia
  Interventions: Drug: Dexamethasone, haloperidol
- dexamethasone + haloperidol 2mg (Active Comparator): dexamethasone 5mg iv during anesthesia induction & haloperidol 2mg iv 30 min before end of anesthesia
  Interventions: Drug: Dexamethasone, haloperidol

INTERVENTIONS:
Drug: Dexamethasone iv injection — Dexamethasone 5mg iv during anesthesia induction
  Arms: dexamethasone
Drug: Dexamethasone, haloperidol — dexamethasone + haloperidol 1mg
  Arms: dexamethasone, haloperiol 1mg
Drug: Dexamethasone, haloperidol — Active Comparator: dexamethasone + haloperidol 2mg
  Arms: dexamethasone + haloperidol 2mg

SUMMARY:
Low-dose haloperidol is known to be effective for the treatment of postoperative nausea and vomiting (PONV). However, precise dose-response studies have not been completed, especially in patients at high risk for PONV who require combination therapy. This study sought to identify the optimal dose of haloperidol that could be combined with dexamethasone without adverse effects in high-risk PONV patients receiving intravenous patient-controlled anesthesia (IV PCA) after gynecological laparoscopic surgery.

DETAILED DESCRIPTION:
Female adults with three established PONV risk factors based on Apfel's score were randomised into one of three study groups. At the end of anaesthesia, groups H0, H1, and H2 were given intravenous (IV) saline, haloperidol 1 mg, and haloperidol 2 mg, respectively. All patients were given dexamethasone during the induction of anaesthesia. The overall early (0-2 h) and late (2-24 h) incidences of nausea, vomiting, rescue anti-emetic administration, pain, and adverse effects (cardiac arrhythmias and extrapyramidal effects) were assessed postoperatively. The sedation score was recorded in the postanaesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II women
* Aged 20 65 years, and scheduled for gynecologic laparoscopic surgery and IV patient-controlled analgesia (PCA) for postoperative pain control.

Exclusion Criteria:

* Known allergy or intolerance to the study drug
* History of cardiac arrhythmia
* Psychiatric illness
* Chronic treatment with a dopamine antagonist
* Use of opioids or steroids within one week of surgery
* Use of antiemetic within 24 hours before the study
* No ability to use the PCA device
* Gastrointestinal, renal, or hepatic disease
* Insulin-dependent diabetes or obesity with a body mass index > 35 kg/m2.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Y.E. Moon, MD, Principal Investigator — associate proffesor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joo J, Park YG, Baek J, Moon YE. Haloperidol dose combined with dexamethasone for PONV prophylaxis in high-risk patients undergoing gynecological laparoscopic surgery: a prospective, randomized, double-blind, dose-response and placebo-controlled study. BMC Anesthesiol. 2015 Jul 8;15:99. doi: 10.1186/s12871-015-0081-1. PMID 26152218

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg
Started | 50 | 50 | 50
Completed | 50 | 49 | 50
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg | Total
Number analyzed (Participants) | 50 | 49 | 50 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 49 | 50 | 149
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 50 | 149
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 50 | 49 | 50 | 149

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Nausea and Vomiting
Description: incidence of nausea, vomiting and requirement for rescue antiemetics
Time Frame: postoperative 24 hours
Measure: Number; unit: participants
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg
Number analyzed (Participants) | 50 | 49 | 50
participants | 21 | 11 | 10

2. Secondary Outcome: Incidence of Extrapyramidal Symptoms
Time Frame: postoperative 24 hours
Measure: Number; unit: participants
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg
Number analyzed (Participants) | 50 | 49 | 50
participants | 0 | 0 | 0

3. Secondary Outcome: Incidence of Cardiac Arrhythmia
Description: cardiac arrhythmia on continuous standard lead EKG monitoring
Time Frame: postoperative 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg
Number analyzed (Participants) | 50 | 49 | 50
Participants | 0 | 0 | 0

4. Secondary Outcome: Sedation Change in Recovery Room
Description: measurement of sedation change using a visual analogue scale (visual analogue scale; the minimum: 0 = widely awake and the maximum: 10 = maximally asleep)
Time Frame: postoperative 30, 60, 90, and 120 min
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg
Number analyzed (Participants) | 50 | 49 | 50
score on a scale
  postoperative 30 min | 4.6 (1.3) | 4.7 (1.0) | 5.5 (1.1)
  postoperative 60 min | 4.4 (1.3) | 4.4 (1.0) | 5.0 (1.0)
  postoperative 90 min | 3.5 (1.4) | 4.0 (1.2) | 4.7 (0.9)
  postoperative 120 min | 3.0 (1.0) | 3.2 (1.1) | 4.3 (1.3)

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Dexamethasone, Haloperiol 1mg | Dexamethasone + Haloperidol 2mg
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No